CLINICAL TRIAL: NCT05727319
Title: Advances in Imaging to Assess Response in Pancreatic Cancer (AIR-PANC): a Single Centre Feasibility Study
Brief Title: Advances in Imaging to Assess Response in Pancreatic Cancer (AIR-PANC)
Acronym: AIR-PANC
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN21ON523
Record Dates: First submitted 2023-01-11; First posted 2023-02-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: PDAC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample and biopsy tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to determine the feasibility of acquiring serial MRI images for longitudinal analysis in pancreatic ductal adenocarcinoma (PDAC) patients. The main question it aims to answer:

Is it feasible to acquire baseline and repeat MR images in Radiotherapy treatment position?

DETAILED DESCRIPTION:
PDAC is one of the leading causes of cancer deaths in the UK, with the number of deaths resembling the number of new cases each year. Long term survival is poor, with around 3% of patients alive at 5 years, reducing to 1% at 10 years. Outcomes have shown minor improvement over the past few decades, with little impact in survival being achieved. This is a worldwide problem, with pancreatic cancer being 7th cause of cancer death.

Although progress has been made in terms of assessing the molecular profiling of pancreatic cancer, there has been little progress in some of the clinical aspects e.g. optimal radiological assessment to stratify patients. Currently imaging criteria following neo-adjuvant treatment has been shown to be sub-optimal in accurately defining response to treatment, which may prevent patients from receiving the treatment that gives them the best outcomes. The emerging paradigm in using pre-operative treatment (chemotherapy +/- RT) to improve outcomes for patients is likely to become the standard of care, increasing the need for advanced imaging assessments that accurately stratify patients by enhancing what is currently assessable on morphological images.

Quantified imaging biomarkers (QIMB) and radiomics are a highly promising area of RT research which will enhance the future direction of personalised treatment. Groups have used said research to examine tumour response; predict toxicity; and adapt RT for some anatomical sites. However, this area of research is particularly challenging in the abdomen, where many uncertainties exist, e.g. motion of pancreas and organs at risk; and poor image quality due to motion artefacts on imaging. New promising data is emerging from centres where patients are being treated with MR guided radiotherapy (MRgRT) systems. These include serial image analysis using delta radiomics that can predict early response in tumour; and feasibility of acquiring functional MR throughout treatment that shows apparent diffusion coefficient (ADC) change in tumour and a correlation to response. Very little work has been done to measure ADC changes during RT and this is where potential to adapt RT lies.

Diffusion MRI (dMRI) allows increased monitoring of functional changes during or post RT by providing information on the biological characteristics of tissue. Recent data even shows promise in the correlation of treatment outcome to ADC measured or compared pre and post RT, by correlating change in ADC to pathologic response; as a tool to predict patients likely to have a successful R0 resection; and in predicting patients who will not respond to CRT and may require a different disease management.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed localised PDAC -as determined by the West of Scotland Hepato-Pancreatobiliary (HPB) MDT
* Scheduled to undergo RT +/- chemotherapy
* 18 years of age or older
* Measurable disease on imaging
* Able to give written informed consent
* Patients willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* Distant metastatic disease
* Other severe or uncontrolled systemic disease or evidence of any other significant disorder or lab finding that makes it undesirable for the patient to participate in the study, as determined by the treating physician.
* History of physical or psychiatric disorder that would prevent informed consent and compliance with protocol
* Major surgery within 28 days prior to trial entry
* Any contraindication to MR
* MRI unsafe implants, ferrous metal in the body, insufficient information on previous surgeries, MRI conditional implants where the conditions cannot be met (e.g. pacemakers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PDAC patients scheduled to undergo RT +/- chemotherapy at the BWOSCC will be recruited where eligibility criteria are met. These patients will have confirmed pancreatic ductal adenocarcinoma (PDAC) which is locally advanced pancreatic cancer (LAPC), or borderline resectable pancreatic cancer (BRPC). Study duration is expected to be 18 months from first patient recruited.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Reproduciblity | 18 months
  The proportion of patients who have successfully completed acquisition of a baseline and week 1 repeat scans
Volumetric and functional feasibility | 18 months
  The proportion of patients where volumetric and functional measurements are reproducible between baseline and repeat scans
Region of interest quantifiability | 18 months
  The proportion of patients where a region of interest can be created and quantified imaging parameters (e.g. ADC) can be extracted on baseline and repeat imaging

SECONDARY OUTCOMES:
Image parameter extraction | 18 months
  The proportion of patients where a region of interest (ROI) can be created and quantified imaging parameters (e.g. ADC) can be extracted on baseline and repeat imaging
Morphological data | 18 months
  The proportion of patients where change in ADC pre and post RT correlate to RECIST from SOC to follow up
Reproducibility of motion corrected/gated image acquisition | 18 months
  The proportion of patients where key features can be tested on larger data sets

OTHER OUTCOMES:
Metabolic changes | 18 months
  The proportion of patients with RT induced metabolic changes that are predictive of outcomes in PDAC
Translational | 18 months
  The proportion of patients where transcriptomic subtypes of pancreatic cancer to baseline dMRI and changes of dMRI post RT as a discovery biomarker analysis of response prediction
Prognostic tool discernment | 18 months
  The proportion of patients where the systemic metabolic fingerprint of the tumour can be used as a prognostic tool to discern response to radiotherapy
Characterisation | 18 months
  The proportion of patients where the processing of FFPE tissue samples with the Human Whole Transcrtiptome TempO-seq assay for 10 patients can be successfully collected and analysed

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Duffton, Study Chair — Chief Investigator
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom